CLINICAL TRIAL: NCT01346787
Title: A MULTICENTER, OPEN LABEL PHASE II STUDY OF CARFILZOMIB, CYCLOPHOSPHAMIDE AND DEXAMETHASONE IN NEWLY DIAGNOSED MULTIPLE MYELOMA PATIENTS
Brief Title: Carfilzomib, Cyclophosphamide and Dexamethasone In Newly Diagnosed Multiple Myeloma Patients
Acronym: CCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-506
Record Dates: First submitted 2011-04-19; First posted 2011-05-03 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: carfilzomib; dexamethasone; cyclophosphamide; multiple myeloma; newly diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib Cyclophosphamide Dexamethasone (Experimental): The treatment period includes administration of Carfilzomib Cyclophosphamide Dexamethasone for 9 courses. In order to assess the toxicity of treatment, patients will attend the study centre visits at each scheduled carfilzomib administration. The response will be assessed after each cycle.
  Interventions: Drug: CARFILZOMIB, CYCLOPHOSPHAMIDE, DEXAMETHASONE

INTERVENTIONS:
Drug: CARFILZOMIB, CYCLOPHOSPHAMIDE, DEXAMETHASONE — Patients will start induction treatment with Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15. Low dose Dexamethasone will be given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23. Carfilzomib = 20 mg/m2 IV once daily on days 1, 2, of cycle 1 only followed by 36 mg/ m2 days 8, 9, 15, 16 in cycle 1, then for all subsequent doses 36 mg/ m2 IV once daily on days 1, 2, 8, 9, 15, 16, followed by 13-day rest period (day 17 through 28). Each cycle will be repeated every 28 days for a total of 9 courses. MANTEINANCE PERIOD At the end of induction phase (9 courses), maintenance phase with Carfilzomib alone IV at 36 mg/ m2 IV on days 1, 2, 15, 16 will start, until progression or intolerance. For patients who show evidence of progression during maintenance phase, the frequency of Carfilzomib can be increased to days 1, 2, 8, 9, 15, 16 at the discretion of the investigator, or the patient may be removed from the study

SUMMARY:
The purpose of this study is to determine whether the association of Carfilzomib, Cyclophosphamide and Dexamethasone (CCd) as induction treatment is safe and provides benefits in patients with newly diagnosed Multiple Myeloma (MM).

DETAILED DESCRIPTION:
This protocol is a phase II multicenter, international, non-comparative, open label study designed to jointly assess the safety and the efficacy of the association Carfilzomib with Cyclophosphamide and Dexamethasone (CCd) as induction treatment and Carfilzomib alone as maintenance in newly diagnosed MM patients.

Patients will be evaluated at scheduled visits in up to 4 study periods: pre-treatment, treatment, maintenance and long-term follow-up.

The pre-treatment period includes screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. The screening period includes the availability of inclusion criteria described above.

The treatment period includes administration of Carfilzomib, Cyclophosphamide and Dexamethasone for 9 4-week courses. In order to assess the toxicity of treatment, patients will attend the study centre visits at each scheduled Carfilzomib administration. The response will be assessed after each 4-week cycle.

The maintenance period includes carfilzomib alone on days 1, 2, 15, 16 at 36mg/m2. For patients who show evidence of progression during maintenance phase, the frequency of Carfilzomib can be increased to days 1, 2, 8, 9, 15, 16 at the discretion of the investigator. It will be initiated at the end of the 9th course and will be stopped at progression or intolerance. The median expected duration of the maintenance treatment is approximately 2 years.

The Long Term Follow Up periods will start after development of confirmed Progression Disease, all patients are to be followed for survival during the Long Term Follow Up period every 3 months via telephone or office visit.

Approximately 15 Italian centers and foreign centers will participate to the protocol.

Patients with symptomatic newly diagnosed MM whose age is ≥ 65 years or who are ineligible for autologous stem cell transplantation. Up to 53 patients will be enrolled from different centers.

The duration of the treatment is approximately 9 months. This length of time is required to complete 9 courses of CCd. At the end of the first stage (19 patients), the trial will be temporarily stopped until all 19 patients complete the toxicity and efficacy evaluation (3 cycle): if there are more than 7 responses and less than 8 toxicities, a further group of 34 patients (total=53) will be enrolled. Otherwise, the trial will be definitively stopped or the DSMC will recommend testing other doses of the drugs.

The maintenance period in both phases will start at the end of the 9th course and will be stopped at progression or intolerance. The median expected duration of the maintenance treatment is approximately 2 years. The duration of follow-up from relapse will be approximately 2 years. The occurrence of PD will determine the duration of TTP of each patient. The occurrence of death will determine the duration of overall survival. The first analysis to evaluate safety and efficacy is planned when the 19 patients enrolled in the first stage of the study have completed the third cycle of induction treatment.

The trial will be stopped if there are < 6 responses, or > 9 toxicities or the Data Safety Monitoring Committee recommends testing other doses of the drugs; Otherwise, a further group of 34 patients (total=53) will be enrolled. The final conclusion will be negative if there are ≤ 23/53 responses, or ≥ 20/53 drug-related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of a legally consenting age as defined by local regulations.
* Patient is age ≥ 65 year of age or who are ineligible for autologous stem cell transplantation.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
* Patient is a newly diagnosed MM patient.
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.
* - Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline (day

  1 of the Cycle 1, before study drug administration):
* Platelet count ≥50 x 109/L (≥30 x 109 /L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to drug administration).
* Absolute neutrophil count (ANC) ≥ 1 x 109/L without the use of growth factors.
* Corrected serum calcium ≤14 mg/dL (3.5 mmol/L)
* Alanine transaminase (ALT): ≤ 3 x the ULN.
* Total bilirubin: ≤ 2 x the ULN.
* Calculated or measured creatinine clearance: ≥ 15 mL/minute

Exclusion Criteria:

* - Patients with non-secretory MM, unless serum free light chains are present and the ratio is abnormal.
* Pregnant or lactating females
* Patient has active infectious hepatitis type B or C or HIV.
* Patients with myocardial infarction or unstable angina ≤ 4 months or other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Peripheral neuropathy > CTCAE grade 2 and ≥ grade 2 painful peripheral neuropathy (with the difference being in the exclusion of patients with Grade 2 painful PN).
* Known history of allergy to Capsidol (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to baseline;
* Patient has any other clinically significant illness that would, in the investigator's opinion, increase the patient's risk for toxicity.
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix or breast, or localized prostate cancer of Gleason score <7 with a stable PSA)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Toxicity: Assessment of adverse events will be performed at the end of third cycle according to the National Cancer Institute Common Terminology Criteria of Adverse Events (CTCAE version 4.0) | 4 years
  Toxicity is defined as the first occurrence of a grade 4 hematologic drug-related toxicity excluding anemia, (grade 4 neutropenia must last longer than 3 days and grade 4 thrombocytopenia must last longer than 7 days in order to be considered a toxicity) with the exception of (grade 4 neutropenia > 3 days , or grade 4 thrombocytopenia >7 days duration) or grade 3 non-hematologic drug-related toxicity.
Efficacy will be assessed by considering partial response (PR) following the proposed regimen. Assessment of Partial Response rate will be performed at the end of third cycle according to the criteria of the International Myeloma Working Group. | 4 years

SECONDARY OUTCOMES:
Response rate | 4 years
Duration of Progression Free Survival | 4 years
Time to progression (TTP) | 4 years
Duration of Response (DOR) | 4 years
Duration of Overall Survival | 4 years
Time to next therapy | 4 years
Progressio Free Survival | 4 years
  Relation between responses and Progression Free Survival, in responding and non-responding patients.
β2-microglobulin as prognostic factors | 4 years
  Subgroups analysis on prognostic factors
peripheral neuropathy | 4 years
  Rates of peripheral neuropathy, according to the National Cancer Institute Common Toxicity Criteria (version 4.0)
Progression Free Survival | 4 years
  Effect on Progression Free Survival of maintenance with low dose of Carfilzomib (days 1 and 2 every other week)
C reactive protein as prognostic factors | 4 years
  Subgroups analysis on prognostic factors
cytogenetics as prognostic factors | 4 years
  Subgroups analysis on prognostic factors
microRNA | 4 years
  Subgroups analysis on prognostic factors
gene expression profile | 4 years
  Subgroups analysis on prognostic factors
Overall Survival | 4 years
  Effect on Overall Survival of maintenance with low dose of Carfilzomib (days 1 and 2 every other week)

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (12):
  - IRCCS CROB UOC di Ematologia e trapianto cellule staminali Ospedale Oncologico Regionale, Rionero in Vulture, PZ
  - azienda ospedaliero-universitaria umberto I Clinica di Ematologia, Ancona
  - Policlinico S. Orsola Istituto di Ematologia e Oncologia Medica, Bologna
  - Ospedale Ferrarotto_Reparto di Ematologia, Catania
  - Az.Osp. Di Careggi_Dh ematologia, Florence
  - Istituto Nazionale per lo Studio e la Cura dei Tumori_UO Ematologia_Trapianto di Midollo Osseo Allogenico, Milan
  - Divisione di Ematologia Dipartimento di Medicina Clinica e Sperimentale Università Amedeo Avogadro, Novara
  - Cattedra di ematologia Università La Sapienza, Roma
  - Divisione di Ematologia Ospedale S. Eugenio, Roma
  - S.C.di Oncoematologia, Azienda Ospedaliera S. Maria di Terni, Terni
  - SC Ematologia - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - SSD CLINICAL TRIAL IN ONCOEMATOLOGIA E MIELOMA MULTIPLO - A.O.U. Città della Salute e della Scienza di Torino, Torino
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] Mina R, Bonello F, Petrucci MT, Liberati AM, Conticello C, Ballanti S, Musto P, Olivieri A, Benevolo G, Capra A, Gilestro M, Galieni P, Cavo M, Siniscalchi A, Palumbo A, Montefusco V, Gaidano G, Omede P, Boccadoro M, Bringhen S. Carfilzomib, cyclophosphamide and dexamethasone for newly diagnosed, high-risk myeloma patients not eligible for transplant: a pooled analysis of two studies. Haematologica. 2021 Apr 1;106(4):1079-1085. doi: 10.3324/haematol.2019.243428. PMID 32107329
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Bringhen S, Mina R, Petrucci MT, Gaidano G, Ballanti S, Musto P, Offidani M, Spada S, Benevolo G, Ponticelli E, Galieni P, Cavo M, Di Toritto TC, Di Raimondo F, Montefusco V, Palumbo A, Boccadoro M, Larocca A. Once-weekly versus twice-weekly carfilzomib in patients with newly diagnosed multiple myeloma: a pooled analysis of two phase I/II studies. Haematologica. 2019 Aug;104(8):1640-1647. doi: 10.3324/haematol.2018.208272. Epub 2019 Feb 7. PMID 30733270
- [Derived] Palumbo A, Bringhen S, Mateos MV, Larocca A, Facon T, Kumar SK, Offidani M, McCarthy P, Evangelista A, Lonial S, Zweegman S, Musto P, Terpos E, Belch A, Hajek R, Ludwig H, Stewart AK, Moreau P, Anderson K, Einsele H, Durie BG, Dimopoulos MA, Landgren O, San Miguel JF, Richardson P, Sonneveld P, Rajkumar SV. Geriatric assessment predicts survival and toxicities in elderly myeloma patients: an International Myeloma Working Group report. Blood. 2015 Mar 26;125(13):2068-74. doi: 10.1182/blood-2014-12-615187. Epub 2015 Jan 27. PMID 25628469
- [Derived] Bringhen S, Petrucci MT, Larocca A, Conticello C, Rossi D, Magarotto V, Musto P, Boccadifuoco L, Offidani M, Omede P, Gentilini F, Ciccone G, Benevolo G, Genuardi M, Montefusco V, Oliva S, Caravita T, Tacchetti P, Boccadoro M, Sonneveld P, Palumbo A. Carfilzomib, cyclophosphamide, and dexamethasone in patients with newly diagnosed multiple myeloma: a multicenter, phase 2 study. Blood. 2014 Jul 3;124(1):63-9. doi: 10.1182/blood-2014-03-563759. Epub 2014 May 22. PMID 24855212